CLINICAL TRIAL: NCT02334930
Title: Evaluation of New Biomarkers Predictive of Efficacy Betablockers in PEComa and Vascular Pediatric Tumors
Acronym: PEC-Hem
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2013/34
Record Dates: First submitted 2014-12-22; First posted 2015-01-08 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: PEComa; Hemangioma
Keywords: propranolol; betablocker; angiogenesis
MeSH Terms: conditions — Perivascular Epithelioid Cell Neoplasms; Hemangioma | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients who will have biopsy or surgery for Perivascular epithelioid cell tumor (PEComa) or vascular pediatric tumor (Rapidly Involuting Congenital Hemangioma (RICH), Non Involuting Congenital Hemangioma (NICH), hemangioma or pyogenic granuloma)
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy

SUMMARY:
PEComa is rare tumor affecting particularly patients with Tuberous Sclerosis. Biological similarities were seen between PEComa and infantile hemangioma. Propranolol is highly efficient to treat infantile hemangioma and we believe that this drug can also be useful for the treatment of PEComa.

Purpose : to understand the mechanism of action of propranolol in PEComas and related pediatric vascular lesions and to select possible novel targets of betablockers in vascular tumors related to PEComas by using YAP oncogene activation as a molecular marker

ELIGIBILITY:
Inclusion Criteria:

* patients who will have biopsy or surgery for PEComa or vascular pediatric tumor (RICH, NICH, hemangioma or pyogenic granuloma)
* A free, informed and written consent will be established

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who will have biopsy or surgery for PEComa or vascular pediatric tumor (RICH, NICH, hemangioma or pyogenic granuloma)
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
YAP cellular expression by immunohistochemistry study on collected tissues | At inclusion (day 0)]

SECONDARY OUTCOMES:
Beta adrenergic receptors expression by immunohistochemistry study on collected tissues | At inclusion (day 0)]
Study of Hippo/YAP pathway expression by western-blot, and correlation with propranolol efficacy | At inclusion (day 0)]
Study of MAP/kinases pathway expression by western-blot, and correlation with propranolol efficacy | At inclusion (day 0)]
Study of PKA/AMPc pathway expression by western-blot, and correlation with propranolol efficacy | At inclusion (day 0)]

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France